CLINICAL TRIAL: NCT00083031
Title: Metronomic Chemotherapy With Bevacizumab for Advanced Breast Cancer
Brief Title: Metronomic Low-Dose Cyclophosphamide and Methotrexate With or Without Bevacizumab in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Harold J. Burstein, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-083; P50CA089393 (NIH); P30CA006516 (NIH)
Record Dates: First submitted 2004-05-14; First posted 2004-05-17 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Cyclophosphamide; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A-Bevacizumab (Experimental): * Methotrexate- twice daily on predetermined days per each week per cycle
  * Cyclophosphamide- oral, daily, predetermined dose
  * Bevacizumab- Via IV on predetermined days per cycle
  Interventions: Drug: bevacizumab; Drug: cyclophosphamide; Drug: methotrexate
- Arm B- Without Bevacizumab (Experimental): * Methotrexate- twice daily on predetermined days per each week per cycle
  * Cyclophosphamide- oral, daily, predetermined dose
  Interventions: Drug: cyclophosphamide; Drug: methotrexate

INTERVENTIONS:
Drug: bevacizumab
  Other Names: Avastin
  Arms: Arm A-Bevacizumab
Drug: cyclophosphamide
  Other Names: Cytoxan; Neosar
Drug: methotrexate
  Other Names: Otrexup™; Rasuvo®; Rheumatrex®; Trexall

SUMMARY:
This randomized phase II trial is studying metronomic low-dose cyclophosphamide and methotrexate to see how well they work compared to metronomic low-dose cyclophosphamide, methotrexate, and bevacizumab in treating women with metastatic breast cancer.

DETAILED DESCRIPTION:
This study uses an investigational drug called Bevacizumab. Investigational means that this drug is not approved by the Federal Drug Administration and is still being studied. Bevacizumab is the common name for the commercial drug Avastin. The Bevacizumab used in this trial, however, is for use in research studies only and may be made at locations different from those where Avastin is made. Although some differences may exist, bevacizumab for research use and the commercial drug, Avastin, are manufactured by a similar process, meet similar standards for final product testing, and are expected to be very similar in safety and effectiveness.

The purpose of this study is to find out what effects (good and bad) low-dose continuous chemotherapy (referred to as metronomic chemotherapy) using drugs Cytoxan (also called cyclophosphamide) and methotrexate (CM), with or without bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed invasive breast cancer, with stage IV disease. Patients without pathologic or cytologic confirmation of metastatic disease should have unequivocal evidence of metastasis by physical exam or radiologic study.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan. The protocol will employ the RECIST criteria.
* Prior Therapy:

  * Chemotherapy: early stage breast cancer. Patients may have received prior adjuvant chemotherapy and/or hormonal therapy for early stage breast cancer, including cyclophosphamide-based chemotherapy regimens.
  * Chemotherapy: metastatic breast cancer. Patients may have received 0-1 prior regimens for metastatic breast cancer. No prior oral cyclophosphamideor methotrexate-based therapy for metastatic disease is permitted.
  * Chemotherapy: anthracyclines. Patients without prior anthraycline (in either the metastatic or adjuvant setting) exposure are eligible provided that they do not have visceral (parenchymal lung or liver) metastases. Patients without prior anthracycline-based therapy are expected to have "low volume" tumor burden, deemed appropriate for non-standard chemotherapy in the estimation of the treating clinician.
  * Trastuzumab. Patients with HER2-positive breast tumors must have received prior trastuzumab therapy for advanced disease, or have had recurrence within 12 months of receiving (neo)adjuvant trastuzumab.
  * Radiation therapy. Patients may have received prior radiation therapy in either the metastatic or early stage settings. Radiation therapy may not be administered during the study. Lesions progressing after previous irradiation are measurable; lesions not progressing after previous irradiation are not measurable.
  * Hormonal therapy. Patients with estrogen- or progesterone-receptor positive disease must have received at least one prior hormonal therapy in the adjuvant and/or metastatic setting.

    --- Patients must discontinue chemotherapy and/or hormonal therapy prior to study participation.
  * Concurrent Therapy. Patients may receive concurrent bisphosphonate therapy and/or erythropoietin growth factor support while on study. Patients may not receive other experimental treatments while on study. Bisphosphonate therapy and/or erythropoietin growth factor support therapy may commence at any point on study.
* Patients may not have received prior experimental angiogenesis inhibitors.
* Age ≥18 years.
* Life expectancy greater than 6 months.
* ECOG performance status ≤ 1 (Karnofsky ≥70%; see Appendix B).
* Absence of poorly controlled hypertension (as defined by the treating clinician), proteinuria, prior history of either deep venous or arterial thrombosis, bleeding diatheses (including hemoptysis).
* Radiologic exclusion of brain metastases (because of concern for potential CNS bleeding with therapy). All patients must have a brain CT or MRI no more than 6 weeks prior to enrollment.
* Left ventricular function ≥ 45% as assessed by echocardiogram or nuclear medicine gated study.
* Patients must have normal organ and marrow function as defined below. Labs should be completed within 4 weeks prior to registration.

  * absolute neutrophil count ≥1000/mm3
  * platelets ≥100,000/mm3
  * total bilirubin ≤ 2 x institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤ 4.0 x ULN
  * Alkaline phosphatase ≤ 5.0 x ULN
  * creatinine ≤ 2.0 mg/dl
  * 24 hr urine specimen < 500 mg protein/24 hr

    --- or
  * Protein on urinalysis < 1+
  * PT, PTT ≤ institutional upper limit of normal (ULN)
* Fertility/reproduction. Patients must be neither pregnant nor expect becoming pregnant or conceiving a child while on study. Women of childbearing potential must have a negative pregnancy test. The effects of bevacizumab, methotrexate, and cyclophosphamide on the developing fetus are unknown. For this reason, women of childbearing potential must agree to use adequate contraception prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.
* Exclusion Criteria
* Patients with less than stage IV disease or lack measurable disease.
* Prior therapy that included any of the following:

  * Chemotherapy for metastatic breast cancer. Patients who have received ≥ 2 prior regimens for metastatic breast cancer; or who have received prior oral cyclophosphamide- or methotrexate-based therapy for metastatic disease.
  * Patients who have not recovered from reversible adverse events due to prior treatments.
  * Patients still on hormonal therapy - including LHRH agonist therapy.
* Current use of anticoagulants or chronic aspirin therapy (> 325 mg/day) - excluding low-dose warfarin used for venous access patency (doses of 1 to 2 mg/d.)
* History of grade 3 or 4 allergic reactions attributed to compounds of similar chemical or biologic composition to cyclophosphamide (such as other alkylating agents) or methotrexate (such as other antimetabolites.)
* Patients with recent (within 6 months) arterial thromboembolic events, including transient ischemic attack (TIA), cerebrovascular accident (CVA), unstable angina, or myocardial infarction (MI). Patients with clinically significant peripheral artery disease should also be excluded.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with visceral metastases unless they have previously been treated with an anthraycline-based chemotherapy regimen in either the metastatic or adjuvant setting.
* Patients may not receive other investigational agents while on study.
* Non-healing wounds or major surgical procedures other than for venous access device or diagnostic study are not permitted within 28 days prior to enrollment (because of rare potential risk of delayed wound healing associated with bevacizumab).
* Patients with large or rapidly accumulating pleural or abdominal effusions (based on clinician's judgment) because of the theoretical risk for methotrexate accumulation and related toxicity. --- If a patient's condition is deteriorating, laboratory evaluations should be repeated ≤ 48 hours prior to initiation of therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2003-07 (Actual); Primary Completion 2006-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Disease evaluations occurred every 8 weeks for the first 6 cycles and every 12 weeks thereafter until progression, death or lost-to-follow-up. Patients were followed for ORR up to approximately 1 year.
  ORR is the proportion of patients achieving Complete Response (CR) or Partial Response (PR) based on RECIST 1.0 criteria: CR is complete disappearance of all target lesions; PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. Both require confirmation no fewer than 4 weeks apart. CR/PR assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Disease evaluations occurred every 8 weeks for the first 6 cycles and every 12 weeks thereafter until progression, death or lost-to-follow-up. Patients were followed for PFS up to approximately 1 year.
  PFS based on the Kaplan-Meier method is defined as the time from study entry and documented disease progression (PD) per RECIST 1.0 criteria or death. Patients alive without progression are censored at time of last disease assessment. Per RECIST 1.0 for target lesions, PD is at least a 20% increase in sum LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or appearance of new lesions. For non-target lesions, PD is the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Overall Survival (OS) | Patients were followed until death or lost-to-follow-up. Patients were followed for OS up to approximately 4 years.
  OS based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.

CONTACTS AND LOCATIONS:
Overall Officials: Harold J. Burstein, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Massachusetts General Hosptial, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Sarah Cannon Research Institute, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mayer EL, Tayob N, Ren S, Savoie JJ, Spigel DR, Burris HA 3rd, Ryan PD, Harris LN, Winer EP, Burstein HJ. A randomized phase II study of metronomic cyclophosphamide and methotrexate (CM) with or without bevacizumab in patients with advanced breast cancer. Breast Cancer Res Treat. 2024 Feb;204(1):123-132. doi: 10.1007/s10549-023-07167-9. Epub 2023 Nov 29. PMID 38019444